CLINICAL TRIAL: NCT04491942
Title: A Phase 1 Trial of the ATR Inhibitor BAY 1895344 in Combination With Cisplatin and With Cisplatin Plus Gemcitabine in Advanced Solid Tumors With an Emphasis on Urothelial Carcinoma
Brief Title: Testing the Addition of an Anti-cancer Drug, BAY 1895344, to the Usual Chemotherapy Treatment (Cisplatin, or Cisplatin and Gemcitabine) for Advanced Solid Tumors With Emphasis on Urothelial Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-05428; NCI-2020-05428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-117; 10404 (Other: City of Hope Comprehensive Cancer Center LAO); 10404 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Bile Duct Carcinoma; Advanced Breast Carcinoma; Advanced Cervical Carcinoma; Advanced Endometrial Carcinoma; Advanced Esophageal Carcinoma; Advanced Gastric Carcinoma; Advanced Head and Neck Carcinoma; Advanced Lung Non-Small Cell Carcinoma; Advanced Lung Small Cell Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Ovarian Carcinoma; Advanced Penile Carcinoma; Advanced Pleural Malignant Mesothelioma; Advanced Urothelial Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Distal Bile Duct Cancer AJCC v8; Stage III Intrahepatic Bile Duct Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Penile Cancer AJCC v8; Stage III Pleural Diffuse Malignant Mesothelioma AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Distal Bile Duct Cancer AJCC v8; Stage IV Intrahepatic Bile Duct Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Penile Cancer AJCC v8; Stage IV Pleural Diffuse Malignant Mesothelioma AJCC v8; Triple-Negative Breast Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Penile Neoplasms; Mesothelioma, Malignant; Triple Negative Breast Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; BAY 1895344; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (cisplatin, elimusertib) (Experimental): Patients receive cisplatin IV over 1-2 hours on day 1 and 8, and elimusertib PO QD on days 2 and 9. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Elimusertib
- Arm II (cisplatin, gemcitabine, elimusertib) (Experimental): Patients receive cisplatin IV over 1-2 hours on day 1 and 8, gemcitabine IV over 30 minutes on days 1 and 8, and elimusertib PO QD on days 2 and 9. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Elimusertib; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Elimusertib — Given PO
  Other Names: ATR Inhibitor BAY1895344; ATR Kinase Inhibitor BAY1895344; BAY 1895344; BAY-1895344; BAY1895344
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm II (cisplatin, gemcitabine, elimusertib)

SUMMARY:
This phase I trial identifies the best dose, possible benefits and/or side effects of BAY 1895344 in combination with chemotherapy in treating patients with solid tumors or urothelial cancer that has spread to other places in the body (advanced). BAY 1895344 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cisplatin and gemcitabine are chemotherapy drugs that stop the growth of tumor cells by killing the cells. Combining BAY 1895344 with chemotherapy treatment (cisplatin, or cisplatin and gemcitabine) may be effective for the treatment of advanced solid tumors, including urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety and tolerability of the combination of cisplatin + elimusertib (BAY 1895344) in patients with advanced solid tumors.

II. To establish the safety and tolerability of the combination of cisplatin + gemcitabine + BAY 1895344 in patients with advanced solid tumors with an emphasis on urothelial carcinoma (UC).

III. To establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of cisplatin + BAY 1895344 and cisplatin + gemcitabine + BAY 1895344.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic profile of BAY 1895344 (in the doublet and triplet combinations) and gemcitabine (in the triplet) in combination with cisplatin.

II. To further evaluate the toxicity of the combination of cisplatin + gemcitabine + BAY 1895344 in patients with UC.

III. To evaluate preliminary efficacy observed with cisplatin + BAY 1895344 and cisplatin + gemcitabine + BAY 1895344 in patients with advanced solid tumors, including UC.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation of biomarkers, including deleterious deoxyribonucleic acid (DNA) damage response (DDR) gene alterations and circulating tumor (ct)DNA with responses to therapy using whole exome sequencing (WES) and messenger ribonucleic acid sequencing (RNA seq) analysis of archival formalin fixed paraffin embedded (FFPE) tissue, as well as blood.

II. To correlate drug exposure with response and/or toxicity.

OUTLINE: This is a dose-escalation study of elimusertib. Patients are assigned to 1 of 2 arms.

ARM I (DOUBLET COMBINATION): Patients receive cisplatin intravenously (IV) over 1-2 hours on day 1 and 8, and elimusertib orally (PO) once daily (QD) on days 2 and 9. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM II (TRIPLET COMBINATION): Patients receive cisplatin IV over 1-2 hours on day 1 and 8, gemcitabine IV over 30 minutes on days 1 and 8, and elimusertib PO QD on days 2 and 9. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed advanced solid tumor with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria, for which cisplatin-based therapy would be considered appropriate, including:

  * Non-small cell lung cancer (NSCLC)
  * UC
  * Penile cancer
  * Malignant pleural mesothelioma
  * Small cell lung cancer
  * Biliary tract cancer
  * Esophageal and gastric cancers
  * Ovarian cancer
  * Endometrial cancer
  * Cervical cancer
  * Head and neck cancer
  * Triple-negative breast cancer (Her2/neu-negative, estrogen receptor [ER]/progesterone receptor [PR]-negative breast cancer)
* For the expansion cohort of the triplet combination at MTD/RP2D only:

  * Patients with histologically confirmed advanced or unresectable urothelial carcinoma are eligible
  * The histology should be predominantly urothelial (>= 50% of sample evaluated contains urothelial histology)
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of BAY 1895344 in combination with gemcitabine and cisplatin in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Availability of archival FFPE tissue
* Prior cisplatin exposure of < 300 mg/m^2. Patients with prior cisplatin treatment must have received last cisplatin treatment > 6 months prior to enrollment
* Prior treatment with PARP inhibitors is permitted (such as olaparib, rucaparib, or other experimental inhibitors of PARP administered in a clinical trial)
* Prior immune checkpoint inhibitor therapy is permitted (including anti-programmed cell death protein 1 [PD-1], anti-PD-ligand [L]1 therapy, such as pembrolizumab, nivolumab, avelumab, durvalumab, atezolizumab, or anti-cytotoxic t-lymphocyte protein 4 [CTLA4] therapy such as ipilimumab, or other experimental immune checkpoint pathway inhibitors administered in a clinical trial)
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 9 g/dL
* Neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional upper limit of normal (ULN)
* Creatinine clearance >= 40 mL/min OR glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy; patients with stable brain metastases that are asymptomatic and on a stable dose of steroids are also considered eligible
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional classification. To be eligible for this trial, patients should be class 2B or better
* The effects of BAY 1895344, cisplatin, and gemcitabine on the developing human fetus are unknown. For this reason and because deoxyribonucleic acid (DNA)-damage response inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 6 months after completion of BAY 1895344 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of BAY 1895344 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Life expectancy < 6 weeks by investigator assessment
* Other active malignancy requiring treatment, except for cutaneous malignancies that require resection such as squamous cell carcinoma, basal cell carcinoma, or cutaneous melanoma, and except for prostate cancer if only on androgen deprivation therapy
* Significant peripheral neuropathy (grade 2 or higher by Common Terminology Criteria for Adverse Events [CTCAE])
* Sensorineural hearing loss (grade 2 or higher by CTCAE)
* Must NOT have had prior treatment with ATR inhibitor (prior BAY1895344 or other investigational ATR inhibitors), or current treatment with any other investigational agents
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Patients who have targeted therapies (such as PARP inhibitors) within 2 weeks prior to entering the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 1895344 or other agents used in study
* Patients receiving any medications that are substrates of CYP3A4 with a narrow therapeutic window, or strong inhibitors/inducers of CYP3A4 are ineligible, if they cannot be transferred to alternative medication. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because BAY 1895344 as a DNA-damage response inhibitor, cisplatin, and gemcitabine may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 1895344 breastfeeding should be discontinued if the mother is treated with BAY 1895344 and for 4 months after end of treatment. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 28 days after completion of study treatment
  Toxicities will be tabulated and reported according to dose level, grade, type, cycle, and attribution. Tables will be created to summarize these toxicities and side effects, overall and by cohort. Proportions and associated 95% confidence intervals will be calculated for each cohort separately. Cumulative incidence curves will be used to estimate the proportion of patients who will discontinue therapy for reasons of toxicity or general inability to tolerate the regimen.
Recommended phase 2 dose (RP2D) of BAY 1895344 | Up to 21 days from treatment start date

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter - maximum concentration (Cmax) | Day 2 and day 9 after treatment start date
  Estimated using non-compartmental methods. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters will be reported descriptively for exploratory comparison with historical data (gemcitabine).
PK parameter - area under the concentration-time curve (AUC) | Day 2 and day 9 after treatment start date
  Estimated using non-compartmental methods. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters will be reported descriptively for exploratory comparison with historical data (gemcitabine). The impact of cisplatin on BAY 1895344 exposure will be evaluated by calculation of the AUC ratio of (day 9 / day 2) and testing non-parametrically with a null hypothesis of a ratio = 1.
Deoxyribonucleic acid (DNA) damage repair (DDR) mutations | Up to 2 years
  The association between DDR mutations and responses will be described, with a table outlining patients who achieved by progressive disease, stable disease, partial or complete responses and DDR mutation status.
Response rate | Up to 2 years
  The percent of responders will be calculated and associated exact 95% confidence intervals will be constructed.
Progression-free survival (PFS) | Up to 2 years
  Kaplan-Meier plots will be used to summarize PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (8):
- United States (7):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Informed Consent Form: Informed Consent (Doublet Combination Consent) (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04491942/ICF_000.pdf
  • Informed Consent Form: Informed Consent (Triplet Combination Consent) (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04491942/ICF_001.pdf